CLINICAL TRIAL: NCT01497561
Title: A Randomised, Double-blind, Four-period, Cross-over, Dose Response Trial Investigating the Pharmacodynamics and Pharmacokinetics of Single Doses of Insulin Detemir and NPH Insulin in Subjects With Type 2 Diabetes
Brief Title: Pharmacodynamics and Pharmacokinetics of Insulin Detemir in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1538
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin detemir (Experimental)
  Interventions: Drug: insulin detemir
- insulin NPH (Active Comparator)
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Each subject will be randomly allocated to two dose administrations out of four possible doses. Administrated subcutaneously (s.c., under the skin)
  Arms: insulin detemir
Drug: insulin NPH — Each subject will be randomly allocated to two dose administrations out of four possible doses. Administrated subcutaneously (s.c., under the skin)
  Arms: insulin NPH

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacodynamics and pharmacokinetics of single doses of insulin detemir and insulin NPH in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Subjects treated with insulin for minimum 3 months
* Duration of diabetes for at least 12 months
* Body Mass Index (BMI) below 30 kg/m^2
* HbA1c maximum 10% based on analysis from central laboratory

Exclusion Criteria:

* Current treatment with insulin above 1.2 U/kg/day
* Current treatment with insulin glargine
* Current treatment with drugs known to interfere with glucose metabolism
* Current treatment with oral antidiabetic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve

SECONDARY OUTCOMES:
Maximum glucose infusion rate
Time to maximum glucose
Area under the curve
Maximum concentration
Time to maximum concentration
Insulin clearance
Mean residence time of insulin
Terminal rate constant
Terminal half-life

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Germany

REFERENCES:
- [Result] Liebl A, Prager R, Binz K, Kaiser M, Bergenstal R, Gallwitz B; PREFER Study Group. Comparison of insulin analogue regimens in people with type 2 diabetes mellitus in the PREFER Study: a randomized controlled trial. Diabetes Obes Metab. 2009 Jan;11(1):45-52. doi: 10.1111/j.1463-1326.2008.00915.x. Epub 2008 Jul 17. PMID 18643839
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com